CLINICAL TRIAL: NCT04294693
Title: Total Joint Arthroplasty in a Pediatric Population
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-0306.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Total Joint Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Recent Patients: Subjects that have undergone surgical intervention within the past two years from date of study approval and received a total joint arthroplasty and follow up care with Dr. Nathan Donaldson or Dr. Steven Thorpe in the Orthopedics Institute at Children's Hospital Colorado
- New Patients: Subjects that are scheduled to undergo a total joint arthroplasty and/or receive follow-up care with Dr. Nathan Donaldson or Dr. Steven Thorpe at Children's Hospital Colorado
- Long-term follow up Patients: Subjects that received a total joint arthroplasty for non-solid tumor malignancies before May 1, 2017 and no longer follow-up in clinic with Dr. Nathan Donaldson
- Control Group Patients: Subjects with a clinical relationship to Dr. Nathan Donaldson or Dr. Steven Thorpe at Children's Hospital Colorado to act as a control group for statistical matching of the above populations.

SUMMARY:
The primary purpose of this study is to examine the functional ability and quality of life in those patients who received a total joint arthroplasty (TJA) for reasons other than having a solid tumor at the location of the joint.

DETAILED DESCRIPTION:
Patients who undergo a total knee arthroplasty (TKA) or total hip arthroplasty(THA) for non-solid tumor related reasons, are most often those children who developed osteonecrosis or avascular necrosis(AVN) as a side effect of their therapy for leukemia. Other patients undergo TKA or THA after degeneration of their joints secondary to trauma, infection, rheumatologic conditions, or congenital deformity. While not all cases of injury to the knee or hip result in the need for a joint replacement, the quality of life is believed to be improved in these children, as having a functioning joint without pain is believed to be better for the patients' quality of life than ambulating with a painful and/or partially necrotic joint.

ELIGIBILITY:
Inclusion Criteria: Populations 1,2,3

* Age between 10 years and 25 years
* Undergoing or have undergone total joint arthroplasty at Children's Hospital Colorado for non-solid tumor related reasons
* Treated at Children's Hospital Colorado by Dr. Nathan Donaldson, DO or Dr. Steven Thorpe, MD or previously by Travis Heare, MD

Exclusion Criteria: Populations 1,2,3

* Subjects and/or parents not capable of completing basic questionnaires in English (HRQL data will not be collected from non-English speaking subjects because we do not have access to versions of these questionnaires that have been validated in languages other than English. These patients may be included at a later date when validated questionnaires are available).
* Subjects who underwent hemiarthroplasties, failed rotationplasty to arthroplasty conversions, or joint arthroplasty directly related to a tumor at the location of the joint
* Subjects diagnosed with mucopolysaccharidoses (MPS), pseudorheumatoid chondrodysplasia, or diastrophic dwarfism

Inclusion Criteria: Population 4

* Age between 10 years and 25 years
* Treated at Children's Hospital Colorado by Dr. Nathan Donaldson, DO, or Dr. Steven Thorpe, MD or previously by Travis Heare, MD
* Symptomatic joint pain treated non-invasively via lifestyle modifications, over the counter or prescription pain medication, nerve blocks or steroid injections, and/or physical therapy
* Symptomatic joint pain treated via core decompression surgery at Children's Hospital Colorado by Dr. Nathan Donaldson, DO, or Dr. Steven Thorpe, MD, or previously by Travis Heare, MD

Exclusion Criteria: Population 4

* Patients who underwent a joint arthroplasty directly related to a tumor at the location of the joint at Children's Hospital Colorado. Patients undergoing or have undergone total joint arthroplasty at Children's Hospital Colorado for non-solid tumor related reasons
* Subjects diagnosed with mucopolysaccharidoses (MPS), pseudorheumatoid chondrodysplasia, or diastrophic dwarfism

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Study Population 1. Recent Patients: Subjects that have undergone surgical intervention within the past 2 years from date of study approval & received a total joint arthroplasty & follow up care with Dr. Nathan Donaldson or Dr. Steven Thorpe in the Orthopedics Institute at Children's Hospital Colorado .
  * Study Population 2. New Patients: Subjects that are scheduled to undergo a total joint arthroplasty &/or receive follow-up care with Dr. Nathan Donaldson or Dr. Steven Thorpe at Children's Hospital Colorado .
  * Study Population 3. Long-term follow up Patients: Subjects that received a total joint arthroplasty for non-solid tumor malignancies before 05/01/2017 & no longer follow-up in clinic with Dr. Nathan Donaldson.
  * Study Population 4. Control group Patients: Subjects with a clinical relationship to Dr. Nathan Donaldson or Dr. Steven Thorpe at Children's Hospital Colorado to act as a control group for statistical matching of the above populations.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2050-03 (Estimated); Study Completion 2061-03 (Estimated)

PRIMARY OUTCOMES:
Standard of Care Data (routinely collected in clinic) | 10 years
  Demographic information such as specific diagnoses leading to joint degeneration, age at diagnosis, type of medical treatments leading to need for joint replacement, previous treatments for joint including surgeries, complications, etc.
Research Data: Health Related Quality of Life instrument | 10 years
  1. Short Form-36 version 2 (SF-36v2)
Research Data: Health Related Quality of Life instrument | 10 years
  2. Oxford 12 Questionnaire
Research Data: Health Related Quality of Life instrument | 10 years
  3. Modified Harris Hip Score Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Donaldson, DO, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No